CLINICAL TRIAL: NCT06694181
Title: SAFE AND EXPLAINABLE AI-ENABLED DECISION MAKING FOR PERSONALIZED CLINICAL DECISION SUPPORT
Brief Title: Safe and Explainable AI
Status: Not yet recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 34124
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Artifical Inteligence; Cardiology; Breast Cancer; Sepsis
MeSH Terms: conditions — Breast Neoplasms; Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cardiology: The primary objective in this clinical case scenario is to evaluate an ML model utilizing real-time cardiac telemetry, as well as other clinical, demographic, and imaging structured data sources, among hospitalized, intensive care unit (ICU) patients to predict impending inhospital cardiac arrest, identify potentially reversible causes of cardiac arrest, and predict which patients may have impending cardiac arrest due to shockable rhythms i.e. ventricular tachycardia (VT) or ventricular fibrillation (VF).
  Interventions: Other: AI-PERSONALIZED CLINICAL DECISION SUPPORT
- Oncology - Breast Cancer: The primary objective in this clinical case scenario is to evaluate an ML model utilizing structured and unstructured data from clinical, demographic, and tumor molecular and germline sequencing, among outpatients with cancer, to predict short-term mortality and/or symptom decline. The model for prediction to treatment response in breast cancer patients will be compared with two prognostic tools: 1) Conversation Connect, a previously validated machine learning mortality prediction tool that has been used at the University of Pennsylvania for routine clinical decision support, and 2) the Elixhauser Comorbidity Index, a comorbidity-based prognostic index used commonly in research and risk-adjustment.
  Interventions: Other: AI-PERSONALIZED CLINICAL DECISION SUPPORT
- Sepsis: The primary objective in this clinical case scenario is to develop and evaluate an ML model that utilizes multidmodal clinical data (e.g., structured EHR data such as demographics, laboratory test results, and vital signs; unstructured EHR data including the text of clinical encounter notes and, where available, waveforms from real-time cardiac, hemodynamic, and respiratory monitoring devices) to predict the need for initiation of broad-spectrum antimicrobial therapy for hospitalized patients with sepsis. With a focus on implementable and explainable AI, we will produce well calibrated predictions that are also clinically meaningful at the bedside to aid real-time decision-making about diagnosis and treatment initiation. The model for timely diagnosis and intervention in sepsis will be compared with widely used commercial and open-source sepsis prediction models.
  Interventions: Other: AI-PERSONALIZED CLINICAL DECISION SUPPORT

INTERVENTIONS:
Other: AI-PERSONALIZED CLINICAL DECISION SUPPORT — AI-ENABLED DECISION MAKING FOR PERSONALIZED CLINICAL DECISION SUPPORT

SUMMARY:
While current AI technology is suitable for automating some repetitive clinical tasks, technical challenges remain in solving critical and gainful problems in the domains of patient and disease management. The proposed research seeks to address issues in medical AI, such as integrating medical knowledge effectively, making AI recommendations explainable to clinicians, and establishing safety guarantees.

ELIGIBILITY:
Inclusion Criteria:

Cardiology 18 years of age and older, admitted to any of the Penn Medicine hospitals from 2017 to the present. Sepsis 18 years of age at the time of presentation to an emergency department or admission to any Penn Medicine hospital from July 1, 2017, onward will be eligible as this represents the population at risk for acquiring sepsis Oncology 18 years of age and older with a diagnosis of invasive breast cancer (Stage 1-4) in the Penn Cancer registry

Exclusion Criteria All prediction models will exclude patients under the age of 18 from their patient data sets.

Cardiology Patients whose primary admission diagnosis was cardiac arrest Sepsis Those with pre-existing limitations on life-sustaining therapy will be excluded because their eligibility for sepsis definitions, care received, and outcomes, may be significantly and variably affected by pre-existing limitations on care. Oncology There are no other exclusions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will look at EMR data from cardiac, oncology, and patients at risk for acquiring sepsis.
  Each group has clearly defined inclusion-exclusion criteria. For the machine learning model to predict ventricular arrhythmias and in-hospital cardiac arrest, we will construct patient cohorts consisting of adult (i.e., 18 years of age or older) patients admitted to Sickbay-accessible bed within a Penn Medicine hospital from 2020 to the present as well as patients identified as having experienced cardiac arrest using EHR records.
Sampling Method: Non-Probability Sample
Enrollment: 300000 (Estimated)
Dates: Start 2025-11-29 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Neurosymbolic Learning Algorithms | Prototype and develop new learning algorithms; 18 months. Benchmark and evaluate the learning algorithms; 24 months. Publish research results; 24 months
  Develop and evaluate novel algorithms for training neurosymbolic models. We will develop data- and compute-efficient algorithms for end-to-end training of neurosymbolic models. This task will reduce the burden on clinician experts to provide fine-grained labels on voluminous EHR data.
Explanation Methods | Prototype and develop new explanation algorithms; 18 months. Derive certified guarantees for explanations; 18 months. Benchmark and evaluate the explanation algorithms; 24 months. Extend certificates to new properties and tasks; 30 months. Publ
  We will develop new explainable AI techniques that come with verifiable guarantees. These guarantees will enable trust and transparency in AI at a fundamental level.
Methods for Safety Guarantees | Prototype and develop new rule learning algorithms; 30 months. Scale rule learning algorithms to larger data settings; 36 months. Incorporate new primitives to express complex rules; 36 months. Implement rule learning algorithms on baseline tasks
  We will develop new algorithms that can scalably extract complex logical rules governing safety within the data that have statistical guarantees. These techniques will be rooted in statistical analysis and assist users in identifying out of distribution data and detecting anomalies.

IPD SHARING:
Plan to Share IPD: No